CLINICAL TRIAL: NCT00003354
Title: Conventional Versus Laparoscopic-Assisted Surgery in Colorectal Cancer
Brief Title: Conventional Surgery Compared With Laparoscopic-Assisted Surgery in Treating Patients With Colorectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical Research Council (Other Government)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000066336; MRC-CLASICC; NYCTRU-CLASICC; EU-98014; ISRCTN74883561
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2001-01

CONDITIONS: Colorectal Cancer
Keywords: stage I colon cancer; stage II colon cancer; stage III colon cancer; stage IV colon cancer; stage 0 colon cancer; stage 0 rectal cancer; stage I rectal cancer; stage II rectal cancer; stage III rectal cancer; stage IV rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Laparoscopy

INTERVENTIONS:
Procedure: conventional surgery
Procedure: laparoscopic surgery

SUMMARY:
RATIONALE: Laparoscopic-assisted surgery is a less invasive type of surgery for colorectal cancer and may have fewer side effects and improve recovery. It is not yet known if undergoing conventional surgery is more effective than laparoscopic-assisted surgery for colorectal cancer.

PURPOSE: This randomized phase III trial is studying conventional surgery to see how well it works compared to laparoscopic-assisted surgery in treating patients with colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether longitudinal and circumferential resection margins and lymphatic clearances obtained during laparoscopic surgery are different from those obtained with conventional open surgery in patients with colorectal cancer.
* Compare the patterns of loco-regional or distant metastatic spread after these two surgical methods in these patients.
* Compare the morbidity and mortality rates in these patients after these two surgical methods, particularly in terms of the technical or thromboembolic complications that may develop as a consequence of prolonged pneumoperitoneum.
* Compare the disease-free or overall survival of these patients after these two operative procedures.
* Determine, in those patients in whom laparoscopic surgery fails, which investigatory modalities are appropriate for providing pre-operative indications that a patient is an inappropriate candidate for laparoscopic dissection.
* Compare the differences in quality of life between the two operative procedures, particularly in patients with advanced disease.

OUTLINE: This is a randomized, multicenter study.

Patients undergo laparoscopic surgery or conventional open surgery.

Patients are followed at 1 and 3 months following surgery, then every 3 months for the first year, every 4 months for the second year, and then every 6 months thereafter.

PROJECTED ACCRUAL: Approximately 1,200 patients will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed colorectal cancer
* Must be suitable for elective surgical resection by right hemicolectomy, left hemicolectomy, sigmoid colectomy, anterior resection or abdomino-perineal resection
* No adenocarcinoma of the transverse colon
* No synchronous multiple adenocarcinomas

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Pulmonary:

* No contraindication to pneumoperitoneum such as severe cardio-respiratory disease

Other:

* No acute intestinal obstruction
* No prior malignancy within the past 5 years, except basal cell carcinoma, carcinoma in situ of the cervix, or prostate cancer
* Not pregnant
* No gastrointestinal disease that requires surgical intervention, e.g., Crohn's disease, chronic ulcerative disease, familial polyposis

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified
* Adjuvant chemotherapy allowed

Endocrine therapy:

* Not specified

Radiotherapy:

* Preoperative radiotherapy must be administered before randomization into this trial
* Adjuvant radiotherapy allowed

Surgery:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 1996-07; Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: P.J. Guillou, MD, Study Chair — Leeds Cancer Centre at St. James's University Hospital
Locations (13):
- United Kingdom (13):
  - Saxon Clinic, Bucks, England
  - Castle Hill Hospital, Cottingham, England
  - Leeds General Infirmary at Leeds Teaching Hospital NHS Trust, Leeds, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Royal Liverpool and Broadgreen Hospitals, Liverpool, England
  - Imperial College School of Medicine at St. Mary's, London, England
  - Newcastle Upon Tyne Hospitals NHS Trust, Newcastle upon Tyne, England
  - Queen's Medical Centre, Nottingham, England
  - Salford Royal Hospitals NHS Trust, Salford, England
  - Airedale General Hospital, West Yorkshire, England
  - Ninewells Hospital and Medical School, Dundee, Scotland
  - Royal Infirmary of Edinburgh at Little France, Edinburgh, Scotland
  - University Hospital of Wales, Cardiff, Wales

REFERENCES:
- [Result] Guillou PJ, Quirke P, Thorpe H, Walker J, Jayne DG, Smith AM, Heath RM, Brown JM; MRC CLASICC trial group. Short-term endpoints of conventional versus laparoscopic-assisted surgery in patients with colorectal cancer (MRC CLASICC trial): multicentre, randomised controlled trial. Lancet. 2005 May 14-20;365(9472):1718-26. doi: 10.1016/S0140-6736(05)66545-2. PMID 15894098
- [Result] Jayne DG, Brown JM, Thorpe H, Walker J, Quirke P, Guillou PJ. Bladder and sexual function following resection for rectal cancer in a randomized clinical trial of laparoscopic versus open technique. Br J Surg. 2005 Sep;92(9):1124-32. doi: 10.1002/bjs.4989. PMID 15997446
- [Result] Jayne DG, Guillou PJ, Thorpe H, Quirke P, Copeland J, Smith AM, Heath RM, Brown JM; UK MRC CLASICC Trial Group. Randomized trial of laparoscopic-assisted resection of colorectal carcinoma: 3-year results of the UK MRC CLASICC Trial Group. J Clin Oncol. 2007 Jul 20;25(21):3061-8. doi: 10.1200/JCO.2006.09.7758. PMID 17634484
- [Result] Jayne DG, Thorpe HC, Copeland J, Quirke P, Brown JM, Guillou PJ. Five-year follow-up of the Medical Research Council CLASICC trial of laparoscopically assisted versus open surgery for colorectal cancer. Br J Surg. 2010 Nov;97(11):1638-45. doi: 10.1002/bjs.7160. PMID 20629110
- [Result] Taylor GW, Jayne DG, Brown SR, Thorpe H, Brown JM, Dewberry SC, Parker MC, Guillou PJ. Adhesions and incisional hernias following laparoscopic versus open surgery for colorectal cancer in the CLASICC trial. Br J Surg. 2010 Jan;97(1):70-8. doi: 10.1002/bjs.6742. PMID 20013936